CLINICAL TRIAL: NCT03787966
Title: Attenuating Cancer Treatment-related Toxicity in Oncology Patients With a Tailored Physical Exercise Program: Study Protocol of the ATOPE Trial in Women Recently Diagnosed With Breast Cancer
Brief Title: Attenuating Cancer Treatment-related Toxicity in Oncology Patients With a Tailored Physical Exercise Program
Acronym: ATOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Irene Cantarero Villanueva, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATOPE18
Record Dates: First submitted 2018-12-14; First posted 2018-12-27 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Breast Neoplasms
Keywords: Breast neoplasm; Breast cancer; therapeutic exercise; cardiotoxicity; muscle toxicity
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATOPE-B (Experimental): An adapted therapeutic exercise program performed before medical treatment. 18 bouts of 1'5 hours multimodal components: aerobic, strength and fascial release exercises. Bout frequency will be adapted to the recovery status of each patient (heart rate variability training parameters and patient perception).
  Interventions: Other: ATOPE-B
- ATOPE-I (Active Comparator): An adapted therapeutic exercise program performed during medical treatment. 18 bouts of 1'5 hours multimodal components: aerobic, strength and fascial release exercises. Bout frequency will be adapted to the recovery status of each patient (heart rate variability training parameters and patient perception).
  Interventions: Other: ATOPE-I

INTERVENTIONS:
Other: ATOPE-B — Patients will perform therapeutic exercise before medical treatment and will follow the usual care after medical treatment.
  Other Names: Therapeutic exercise before medical treatment
  Arms: ATOPE-B
Other: ATOPE-I — Patients will follow usual care before medical treatment and will perform therapeutic exercise after medical treatment.
  Other Names: Therapeutic exercise during medical treatment
  Arms: ATOPE-I

SUMMARY:
The aim of this study is to determine if therapeutic exercise before anticancer treatment will mitigate the onset or extent of cardiotoxicity comparing to therapeutic exercise performed during anticancer treatment.

DETAILED DESCRIPTION:
The positive relationship between physical exercise and cancer is widely justified in the literature, but an emerging research line warns of its capacity to improve the effectiveness and reduce the toxicity of cancer treatment (responsible for the appearance of side effects and comorbidities), that overload the health care system. To date, there is a lack of knowledge in different subjects: the possibility of implementing individualized exercise programs in clinical environment to mitigate the side effects of cancer treatment; the best moment in natural history of the disease to perform therapeutic exercise; and a tailored dose of exercise that maximizes its benefits.

In this context, the present study will evaluate the effects of a therapeutic exercise program conducted previously at the beginning of the cancer treatment, in the treatments' toxicity against the same program conducted during cancer treatments in women with breast cancer, and its positive effects on both clinical and biological variables and their possible impact on disease-free survival.

This study will be conducted in 3 phases with 110 participants in total: phase 1: a pilot study be carried out to check the feasibility of the proposed physical exercise program; phase 2: to test the effectiveness of the program ATOPE performed prior to surgical medical treatment against the same made during treatment, with a randomized controlled clinical trial; and phase 3: in which it will be integrated into the health service and a larger project will be requested at the international level.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Breast cancer diagnosis I-III stage
* On the waiting list to anticancer medical treatment (at least surgery, chemotherapy and radiotherapy.
* If they meet other criteria which predisposes to higher toxicity.
* Have signed informed consent.
* Have medical clearance for participation.

Exclusion Criteria:

* Patient underwent previous cancer treatments.
* Patients were previously diagnosed with cancer.
* Pregnant patients.
* Patients performing other type of therapeutic exercise at diagnosis time with an intake >or = to 150 moderate-intensity or 75 min of vigorous-intensity a day.
* Therapeutic exercise practice not recommended because psychiatric or cognitive disorders or cute or chronic condition that prevents exercise (advanced lung disease, oxygen requirement, stenosis >70%, metastasis etc.).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | Participants will be followed over 12 months
  To assess cardiac toxicity by echocardiography

SECONDARY OUTCOMES:
Cardiovascular events | Participants will be followed over 12 months
  Number of cardiovascular events registered in a diary
Resting heart rate | Participants will be followed over 12 months
  To assess cardiac function by a Holter
Heart Rate variability | Participants will be followed over 12 months
  To assess cardiac autonomic system balance by a Holter
Muscle loss | Participants will be followed over 12 months
  To assess muscle mass loss by Inbody
Quality of life with the Quality of Life Questionnaire (QLQ)-C30 | Participants will be followed over 12 months
  With the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0. It is used to asses quality of life. It contains 30 items with both multi-item scales and single-item measures. Values are assigned between 1 and 4 (1: not at all, 2: a little, 3: enough, 4: a lot) according to the patient's responses to the item, only in items 29 and 30 evaluate with a score of 1 to 7 (1: lousy, 7: excellent). The scores obtained are standardized and a score between 0 and 100 is obtained, which determines the level of cancer impact on the patient of each of the scales. The high values in the scales of global health and function state indicate a better CV, while in the scale of symptoms it would indicate a decrease in CV since it indicates the presence of symptoms associated with cancer.
Quality of life with the Quality of life Questionnaire (QLQ- BR23) a specific module. | Participants will be followed over 12 months but will not be assessed in baseline
  European Organization for Research and Treatment of Cancer Breast Cancer-Specific Quality of Life Questionnaire (EORTC QLQ-BR23). It is a breast cancer module of EORTC QLQ-C30. This module contains 23 items assessing symptoms and side effects related to different treatment modalities, body image, sexuality, and future perspective. After the scoring procedures for the QLQ-C30, all scale and single-item scores are linearly transformed to a 0 to 100 scale. For the functional scales and single items (ie, body image, sexuality, and future perspective), higher scores represent a better level of functioning. For the symptom scales and single item, a higher score represents a higher level of symptoms.
Chemotherapy regimen | Participants will be followed over 12 months
  type of chemotherapy agent used and number of sessions.
Chemotherapy doses modifications | Participants will be followed over 12 months
  delay of doses or reduction, total doses received from the total expected.
Early session termination. | Participants will be followed over 12 months
  Patient stopped receiving chemotherapy before last >=1 sessions.
Missing bouts due to adverse effects of chemotherapy | Participants will be followed over 12 months
  Adverse effects of chemotherapy treatment and if it was interrupted (>=3 missing consecutive bouts of exercise)
Number of hospitalizations. | Participants will be followed over 12 months
Therapeutic exercise bout modification | Participants will be followed over 12 months
  >=1 bout that required a dose modification during the program and number of bouts modified in total.
Time to treatment failure | Participants will be followed over 12 months
  days from the start to the end of chemotherapy, if it was terminated for toxicity and/or tumor progression.
Program adverse effects reported by the participants. | Participants will be followed over 12 months
  Frequency of serious and non-serious events occurring during program.
Functional capacity | Participants will be followed over 12 months
  assessed by the 6-Minute Walking Test
Handgrip strength | Participants will be followed over 12 months
  assessed by a digital dynamometer: TKK 5101 Grip-D; Takey, Tokyo, Japan
Shoulder strength | Participants will be followed over 12 months
  assessed by an isokinetic test with an isokinetic dynamometer (HUMAC NORM)
Lower limb strength | Participants will be followed over 12 months
  assessed by an isokinetic test with an isokinetic dynamometer (HUMAC NORM)
Abdominal strength | Participants will be followed over 12 months
  assessed by an isokinetic test with an isokinetic dynamometer (HUMAC NORM)
Flexibility | Participants will be followed over 12 months
  assessed by the Modified sit-and-reach test
Waist and hip circumferences | Participants will be followed over 12 months
  assessed by an inelastic tape
Body composition | Participants will be followed over 12 months
  assessed by the InBody
Oxidative stress | Participants will be followed over 12 months
  Thiobarbituric acid reactive substances (TBARS)
Oxidative stress | Participants will be followed over 12 months
  carbonyls and 8-hydroxy-2' -deoxyguanosine (8-OHdG)
Inmune function | Participants will be followed over 12 months
  Number of lymphocytes: (cluster of differentiation (CD) 8 and 4 and regulatory T lymphocytes)
inflammation | Participants will be followed over 12 months
  C-reactive protein (CRP)
inflammation | Participants will be followed over 12 months
  interleukin (IL) 6 and 10
inflammation | Participants will be followed over 12 months
  tumor necrosis factor (TNF) alpha
inflammation | Participants will be followed over 12 months
  insulin-like growth factor 1 (IGF-1)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Cantarero-Villanueva, PhD, Principal Investigator — Physical Therapy Deparment, Faculty of Health Sciences, University of Granada
Locations (1):
- University of Granada, Granada, Spain

REFERENCES:
- [Derived] Postigo-Martin P, Gil-Gutierrez R, Moreno-Gutierrez S, Lopez-Garzon M, Gonzalez-Santos A, Arroyo-Morales M, Cantarero-Villanueva I. mHealth system (ATOPE+) to support exercise prescription in breast cancer survivors: a reliability and validity, cross-sectional observational study (ATOPE study). Sci Rep. 2022 Sep 8;12(1):15217. doi: 10.1038/s41598-022-18706-7. PMID 36076044
- [Derived] Postigo-Martin P, Penafiel-Burkhardt R, Gallart-Aragon T, Alcaide-Lucena M, Artacho-Cordon F, Galiano-Castillo N, Fernandez-Lao C, Martin-Martin L, Lozano-Lozano M, Ruiz-Vozmediano J, Moreno-Gutierrez S, Illescas-Montes R, Arroyo-Morales M, Cantarero-Villanueva I. Attenuating Treatment-Related Cardiotoxicity in Women Recently Diagnosed With Breast Cancer via a Tailored Therapeutic Exercise Program: Protocol of the ATOPE Trial. Phys Ther. 2021 Mar 3;101(3):pzab014. doi: 10.1093/ptj/pzab014. PMID 33528004